CLINICAL TRIAL: NCT04616807
Title: An Observational Study to Describe the Long-term Safety and Effectiveness of Namuscla in the Symptomatic Management of Myotonia in Adult Patients With Non-dystrophic Myotonic Disorders
Brief Title: An Observational Study in Adult Patients With Non-dystrophic Myotonic Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUP/MEX/2018/001
Record Dates: First submitted 2020-10-23; First posted 2020-11-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Mexiletine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mexiletine — Observational Study
  Other Names: Namuscla ™

SUMMARY:
This is a non-interventional, prospective, observational, multicentre study to evaluate the long-term safety and effectiveness of Namuscla in adult patients with NDM.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, observational, multicentre study to evaluate the long-term safety and effectiveness of Namuscla in adult patients with NDM. Namuscla should be prescribed as per the approved Summary of Product Characteristics (SmPC).

Adult patients with non-dystrophic myotonic disorders who have been prescribed Namuscla by the treating physician, and who meet the eligibility criteria will be enrolled in this study.

This includes:

* Patients newly initiated on Namuscla for the treatment of NDM (newly exposed)
* Patients already on Namuscla/ mexiletine at enrolment - For patients receiving mexiletine other than Namuscla, only those who switch to Namuscla will be included in the study.

Patients already being treated with Namuscla/ mexiletine at the time of enrolment will be considered for enrolment provided they meet the eligibility criteria.

The study will be initiated at specialized centres for the treatment of myotonic disorders ("reference centres") in the United Kingdom (UK), France, and Germany, depending on availability of Namuscla in the specific country. Depending on the enrolment and marketing status (availability) of Namuscla in other countries in the EU, inclusion of additional sites in other countries will be considered.

The study population will comprise patients who are diagnosed with non-dystrophic myotonic disorders and considered suitable candidates for the treatment by Namuscla by the investigators according to the approved SmPC. Patients will be enrolled over an approximate 2-year enrolment period and will be followed-up on-treatment for up to 3 years. Each enrolled patient will be observed for 3 years or until discontinuation (if discontinued early).

For all enrolled patients, the baseline would be the latest data available at the enrolment visit.

For the patients already on Namuscla, cumulative data (data related previous exposure as well as current data) will be collected for adverse events (AEs) on Namuscla treatment.

No drug will be supplied for this study; patients will receive medicines through local standard practices. All evaluations and investigations during the study will be performed according to the routine clinical practices and discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male or female patients with non-dystrophic myotonic disorders planned to be started on Namuscla according to the approved SmPC
2. Patients already receiving Namuscla/mexiletine for the treatment of NDM; (for patients on mexiletine other than Namuscla, only those who switch to Namuscla will be enrolled).
3. Patients who understand and are willing to provide informed consent.

Exclusion Criteria:

1. Patients who are enrolled or participating in any other clinical trial for an investigational product. -
2. Hypersensitivity to mexiletine, or to any of the excipients of Namuscla, or hypersensitivity to any local anaesthetic
3. Ventricular tachyarrhythmia
4. Atrial tachyarrhythmia, fibrillation or flutter
5. Complete heart block (ie, third-degree atrioventricular block) or any heart block susceptible to evolve to complete heart block (first-degree atrioventricular block with markedly prolonged PR interval (≥ 240 ms) and/or wide QRS complex (≥ 120 ms), second-degree atrioventricular block, bundle branch block, bifascicular and trifascicular block),
6. Myocardial infarction (acute or past), or abnormal Q-waves
7. Symptomatic coronary artery disease
8. Heart failure with reduced ejection fraction <50%
9. Sinus node dysfunction (including sinus rate < 50 bpm)
10. Patients receiving drugs that can induce torsades de pointes
11. Patients receiving medicinal products with narrow therapeutic index (ie, theophylline, tizanidine, digoxin, lithium, phenytoin or warfarin)
12. Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will target the enrolment of 50 patients who are treated with Namuscla.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-01-24 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1 Proportion of patients with treatment-emergent AEs | Approximately 3 years
  Proportion of patients with treatment-emergent AEs ([TEAEs], including SAEs) from study enrolment to 6, 12, 24 and 36 months on Namuscla
Primary Outcome 2 Proportion of patients requiring dose reduction or treatment discontinuation | Approximately 3 years
  Proportion of patients requiring dose reduction or treatment discontinuation due to AEs (including SAEs).

SECONDARY OUTCOMES:
Secondary Outcome Proportion of patients with AEs /SAEs/ Adverse Event of Special Interest (AESI) | Approximately 3 years
  Proportion of patients with AEs /SAEs/ Adverse Event of Special Interest (AESI) from study enrolment to 6, 12, 24, and 36 months

CONTACTS AND LOCATIONS:
Locations (6):
- France (2):
  - Hôpital Universitaire de La Pitié Salpêtrière, Paris, Cedex
  - CHRU Lille, Lille
- Germany (2):
  - St. Josef-Hospital Klinikum der Ruhr Universitaet Bochum, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Ulm, Klinik für Neurologie, Ulm
- United Kingdom (2):
  - Institute of Neurology, London, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England